CLINICAL TRIAL: NCT03329768
Title: Evaluation of Peripheral Intravenous Catheter and Urinary Catheters Present on Admission to the "Maladies Infectieuses aiguës" Department.
Brief Title: Evaluation of Medical Device
Status: Completed | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-15; 2016-A00673-48 (Other: IDRCB)
Record Dates: First submitted 2017-10-25; First posted 2017-11-06 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Acute Infectious Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A preliminary study was conducted from 01/26/2015 to 10/26/2015 on 605 patients admitted to MIA with an intravenous and/or a urinary catheter.

the investigators analyzed:

* the demographic characteristics of the patient
* the final diagnosis
* the patient's severity and the patient outcome after discharge from MIA
* the justification of the venous and or a urinary catheter
* the duration of the prescription of the device Evaluation on admission of the need to maintain an intravenous or urinary catheter. Adjusting the prescription in terms of duration or withdrawal of the device in order to limit their complications (lymphangitis, superficial thrombophlebitis, bacteremia related to health care, urinary tract infection).

Hypothesis:

Limit the length of stay and reduce the cost of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an intravenous catheter and/or a urinary catheter.
* Patient is more than 18 years old.
* Patient who accepts to have his medical records reviewed for research.
* Patient with health insurance

Exclusion Criteria:

* Refusal of participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with an intravenous and/or urinary catheter on admission in the department of "Maladies infectieuses aigues" (MIA) Hopital de la Timone AP-HM.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2016-09-28 (Actual); Primary Completion 2020-01-25 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
number of patients with intravenous catheter | 3 YEARS
number of patients with urinary catheter | 3 YEARS

CONTACTS AND LOCATIONS:
Overall Officials: jean-olivier ARNAUD, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France